CLINICAL TRIAL: NCT06046287
Title: Phase IIa Study to Evaluate Daratumumab for Polyneuropathy Associated With MGUS
Brief Title: Daratumumab for Polyneuropathy Associated With MGUS
Acronym: Dara-MGUS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Georgetown University (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005648
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Neuropathy; Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Peripheral Nervous System Diseases; Monoclonal Gammopathy of Undetermined Significance | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab and hyaluronidase-fihj (Experimental)
  Interventions: Drug: Daratumumab and hyaluronidase-fihj

INTERVENTIONS:
Drug: Daratumumab and hyaluronidase-fihj — subucatneous, fixed dose 1800mg combination drug product containing rHuPH20 drug substance (2000 U/mL) and daratumumab drug substance (120 mg/mL) will be administered weekly for the first 8 weeks, and then every 2 weeks from week 9 to week 24.
  Other Names: Darzalex Faspro

SUMMARY:
The goal of this clinical trial is to learn about daratumumab and hyaluronidase-fihj in patients with monoclonal gammopathy of undetermined significant (MGUS) who have been diagnosed with peripheral neuropathy suspected to be cause by paraproteinemia. The main question[s] it aims to answer are:

• how well does this medication help improve MGUS associated peripheral neuropathy

Participants will be asked be asked to get some testing done prior to starting the trial in order for us to assess your nerve damage or peripheral neuropathy. This will include blood tests, a complete neurologic examination, surveys and tests called electromyogram and nerve conduction studies. Participants that qualify for the trial will take DARZALEX FASPRO® once a week for two months, followed by every other week from months 3 to month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent
2. A diagnosis of chronic demyelinating neuropathy according to the European Federation of Neurological Societies/Peripheral Nerve Society guidelines for chronic inflammatory demyelinating polyneuropathy (as determined by neurologist) with concurrent diagnosis of monoclonal gammopathy of undetermined significance (MGUS) with an IgM monoclonal peak (see appendix 8)
3. Peripheral neuropathy associated with anti-MAG >7000 BTU, with EMG/NCS consistent with polyneuropathy.
4. Patients will have to have disability associated with their peripheral neuropathy, with a baseline INCAT Sensory Score (ISS) score ≥4.
5. They must have an ataxia score ≥2 (0 = normal, 1 = slight oscillations, 2 = marked oscillations, 3 = severe ataxia), and/or visual analog pain scale (VAS) >4 (from 0 = no pain to 10 = maximal pain).
6. Must meet MGUS diagnostic criteria as diagnosed using IMWG criteria using the following criteria (see section 1 appendix):

   1. Serum monoclonal protein <30g/L
   2. Clonal bone marrow lymphoplasmacytic/plasma cells <10%
   3. Absence of end-organ damage related to the plasma cell dyscrasia*
7. Serum calcium >0.25 mmol/L (>1mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11mg/dL)
8. Renal insufficiency: creatinine clearance <40 mL per minute or serum creatinine >177mol/L (>2mg/dL)
9. Anemia: hemoglobin value of >20g/L below the lowest limit of normal, or a hemoglobin value <100g/L
10. Bone lesions: one or more osteolytic lesion on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement.
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 3 (see appendix)
12. Adequate bone marrow function:

    * Total WBC count ≥ 1,500/mm3, ANC ≥ 1,000/mm3
    * Hemoglobin (Hb) ≥ 8.0 g/dL,
    * Platelet count ≥ 75,000/mm3.
13. Adequate liver function:

    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN)
    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) > 2.5 is permissible if due to disease.
    * Bilirubin ≤ 2 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin for which > 2 x ULN is an acceptable limit)
14. Adequate renal function: creatinine clearance ≥ 20mL/min.
15. Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
16. Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

1. Documented active multiple myeloma, smoldering myeloma, Waldenstroms macroglobulinemia, non-IgM MGUS, plasma cell leukemia or systemic amyloid light chain amyloidosis
2. Concomitant disorder felt to possibly be related to the etiology of the peripheral neuropathy: diabetes, vitamin deficiency, chronic alcohol consumption, drugs, HCV infection.**
3. Prior or current exposure to any of the following:

   1. To daratumumab and Hyaluronidase-fhj or other anti-CD-38 therapies (unless a re-treatment study)
   2. Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
4. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
5. Moderate or severe persistent asthma within the past 2 years (see Appendix section 1), or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
6. Participant is:

   1. Known history of human immunodeficiency virus (HIV)
   2. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative with antibodies to total hepatitis B core antigen [anti-HBc] with or without the presence of hepatitis B surface antibody [anti-HBs]) must be screed using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of HBV vaccination, do not need to be testing for HBV DNA by PCR.
   3. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as a viremia at least 12 weeks after completion of antiviral therapy).
7. Patients who have implanted deep brain stimulators and vagal nerve stimulators.
8. Clinically significant cardiac disease, including:

   1. Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV) [refer to Appendix section 3]
   2. Uncontrolled cardiac arrhythmia
   3. Patients with external pacing wires or intracardiac catheters
9. If patient is unable to sign informed consent due to any serious medical condition, laboratory abnormality or psychiatric illness
10. If patient is pregnant or breastfeeding, a prisoner, or not yet an adult
11. Any life-threatening illness, medical condition, concomitant active cancer, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
ISS score change | 12 months
  changes from baseline to 12 months in functional assessments ISS score

SECONDARY OUTCOMES:
Functional Assessment change | 3, 6, 9,12 months
  absolute change from baseline in functional assessments using clinical examinations (sensory, reflexive)
Change in nerve conduction studies (NCS) | 3, 6, 9, 12 months
  absolute change from baseline in functional assessments using nerve conduction studies (NCS)
Electromyography (EMG) changes | 12 months
  change from baseline in electromyography (EMG) measured at 12 months
Inflammatory Neuropathy Cause and Treatment (INCAT) changes | 3, 6, 9, 12 months
  Absolute change from baseline in clinician-reported functional measures using the modified Rankin Score, Inflammatory Neuropathy Cause and Treatment (INCAT)
Change in health-related quality of life | 3, 6, 9, and 12 months
  Absolute change from baseline in patient reported health-related quality of life (HRQOL) outcomes, assessed by the 36-item Short Form Health Survey (SF-36) measure.
Change in immunofixation (IFE) | 3, 6, 9, and 12 months
  Absolute change from baseline in immunofixation (IFE),
Change in immunoglobulin concentration | 3, 6, 9, and 12 months
  Absolute change from baseline in immunoglobulin concentration
Change in serum protein electrophoresis (SPEP) | 3, 6, 9, and 12 months
  Absolute change from baseline in serum protein electrophoresis (SPEP)
Change in anti-MAG titers (serology) | 3, 6, 9, and 12 months
  Absolute change from baseline in anti-MAG titers (serology)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Doucette, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No